CLINICAL TRIAL: NCT03681665
Title: Use of Iterative Reconstruction Method in Ultralow-dose CT for Follow-up of Patients With Intraabdominal Abscess: Comparison With Standard Dose CT
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0413
Record Dates: First submitted 2018-09-17; First posted 2018-09-24 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Abdominal Abscess
MeSH Terms: conditions — Abdominal Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Abscess: Patients group with abdominal abscess
  Interventions: Other: ultralow dose abdominopelvic CT

INTERVENTIONS:
Other: ultralow dose abdominopelvic CT — In the patient cohort with abdominal abscess, ultralow dose abdominopelvic CT will be performed as a follow-up protocol. Ultralow dose CT has approximately 80~90% reduced radiation dose compared to standard dose CT.

SUMMARY:
Increasing radiation exposure by medical examinations is getting more concerns. For optimal medical imaging, reducing radiation exposure with preservation image quality is important. One of the solutions is use of iterative recontruction of CT examination. In this study, the investigators aimed to investigate the clinical feasibility of ultralow dose abdominopelvic CT with iterative reconstruction in patients with intraabdominal abscess. Patients with intrabdominal abscess usually undergo multiple CT examinations to evaluate treatment response. Therefore, ultralow dose CT can reduce unnecessary radiation exposure in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients who underwent standard dose CT for suspected intraabdominal abscess
2. patients who need follow-up CT to evaluate treatment response of abscess 3) Adult patient, 4) patients who agreed this study protocol

Exclusion Criteria:

1. pregnancy
2. patients with poor renal function (GFR < 30 mL/min/1/73m2)
3. Patients who have allergy to CT contrast media
4. Patients who are not cooperative (e.g., dementia)

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected abdominal abscess from a tertiary care clinic.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Score of subjective image quality of CT image | 1 month
  Score of subjective image quality of CT images consists of overall subjective image quality, noise, diagnostic ability, and artifact.

SECONDARY OUTCOMES:
Effective radiation dose: CTDIvol(volume CT dose index), DLP(dose length product), effective dose(DLPx0.015) | 1 month
  Effective radiation dose between standard dose CT and ultra-low dose CT will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No